CLINICAL TRIAL: NCT02086708
Title: Sonoelastography: Ultrasound Method to Measure Fibrosis of the Liver in Children
Brief Title: Ultrasound Method to Measure Fibrosis of the Liver in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The technology showed rapid acceptance in the general population and we halted our feasibility demonstration study.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Uzma Shah, MD, Associate Professor in Pediatrics, Massachusetts General Hospital for Children, Harvard Medi, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010P000705
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Liver Disease; Non-Alcoholic Fatty Liver Disease; HCV Coinfection; HBV; Drug-Induced Liver Injury
Keywords: Sonoelastography,; Diffuse liver disease,; chronic liver disease,; NASH,; NAFLD,; Elevated Transaminases,; Liver Biopsy,; Fibrosis,; METAVIR
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Chemical and Drug Induced Liver Injury; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Shear Wave Sonoelastography, Fibrosis stage (Experimental): Shear Wave sonoelastography is performed on patients who are scheduled for a non-focal liver biopsy.
  Interventions: Device: Shear Wave sonoelastography

INTERVENTIONS:
Device: Shear Wave sonoelastography — Shear Wave Sonoelastography as a ultrasound technique to measure liver fibrosis is performed on patients scheduled for non-focal liver biopsy. Results are compared with pathological score of fibrosis from liver biopsy.
  Other Names: Supersonic Aixplorer

SUMMARY:
HYPOTHESIS: The investigators hypothesize that sonoelastography (SE) provide accurate quantitative measurements that can be used to stage liver fibrosis in pediatric patients with chronic liver disease.

Specific Aims:

To measure liver stiffness with sonoelastography in pediatric and adolescents with suspect diffuse liver disease who will undergo nonfocal liver biopsy as part of their routine clinical care.

ELIGIBILITY:
Inclusion criteria:

* Patients scheduled for random liver biopsy for routine staging of liver fibrosis
* Pediatric patients patients (ages 1-21)
* Girls or boys
* Suspected liver disease
* Consent to participate in the study

Exclusion criteria:

* Pregnancy
* Acute illness/cognitive impairment resulting in inability to cooperate with ultrasound
* Patients that do not consent to ultrasound guided liver biopsy.
* Contraindications to liver biopsy (e.g. low platelets defined as a platelet count of less than 50,000, and hemophilia/coagulopathy as an INR higher than 1.5.)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uzma Shah, MD, FAAP, Principal Investigator — Massachusetss General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dhyani M, Gee MS, Misdraji J, Israel EJ, Shah U, Samir AE. Feasibility study for assessing liver fibrosis in paediatric and adolescent patients using real-time shear wave elastography. J Med Imaging Radiat Oncol. 2015 Dec;59(6):687-94; quiz 751. doi: 10.1111/1754-9485.12388. Epub 2015 Oct 27. PMID 26503488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. Patients scheduled for Liver Biopsy 2.
Groups:
- Shear Wave Sonoelastography, Fibrosis: Shear Wave sonoelastography is performed on patients who are scheduled for a non-focal liver biopsy.
  Shear Wave sonoelastography: Shear Wave Sonoelastography as a ultrasound technique to measure liver fibrosis is performed on patients scheduled for non-focal liver biopsy. Results are compared with pathological score from liver biopsy.
Period: Overall Study
Arm/Group | Shear Wave Sonoelastography, Fibrosis
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Pediatric and Adolescents
Arm/Group | Shear Wave Sonoelastography, Fibrosis
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: years] — In this study:
  1. The eligibility age range was 1-21 years.
  2. We enrolled subjects with the age with the minimum age value of 1 years and the maximum age value of 21 years.
  years | 17 [1 to 21]
Gender [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Measure Liver Elasticity Value Using Sonoelastography.
Description: Assess liver stiffness as measured by sonoelastography with results of liver biopsy as read by a single-pathologist using the METAVIR criteria (F0-F4).
Time Frame: Day one
Measure: Mean (95% Confidence Interval); unit: kPa
Groups:
- Fibrosis 0: Patients with no Fibrosis on liver biopsy evaluation
- Fibrosis 1: Patients with liver biopsy METAVIR stage 1 on pathology evaluation
- Fibrosis 2: Patients with liver biopsy METAVIR stage 2 on pathology evaluation
- Fibrosis 3: Patients with liver biopsy METAVIR stage 3 on pathology evaluation
- Fibrosis 4: Patients with liver biopsy METAVIR stage 4 on pathology evaluation
Arm/Group | Fibrosis 0 | Fibrosis 1 | Fibrosis 2 | Fibrosis 3 | Fibrosis 4
Number analyzed (Participants) | 10 | 9 | 1 | 3 | 1
kPa | 6.93 [6.33 to 7.44] | 8.33 [6.83 to 10.80] | 6.12 [NA to NA] — For 1 subject, 95% confidence intervals cannot be calculated. | 8.86 [5.7 to 11.4] | 17.85 [NA to NA] — For 1 subject, 95% confidence intervals cannot be calculated.

ADVERSE EVENTS:
Arm/Group | Fibrosis 0 | Fibrosis 1 | Fibrosis 2 | Fibrosis 3 | Fibrosis 4
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/1 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/1 | 0/3 | 0/1

LIMITATIONS AND CAVEATS:
This was meant to be a feasibility study to show that shear-wave sonoelastography can be performed in the pediatric age group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes